CLINICAL TRIAL: NCT04494984
Title: A Stage 2/3, Adaptive, Randomized, Controlled, Double-blind Study to Investigate the Pharmacokinetics, Efficacy and Safety of the Hyperimmune Equine Serum (INM005) in Adult Patients With Moderate to Severe Confirmed SARS-CoV2 Disease.
Brief Title: A Study to Investigate the Pharmacokinetics, Efficacy and Safety of INM005 in Patients With COVID-19.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Inmunova S.A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-INM005-01
Record Dates: First submitted 2020-07-29; First posted 2020-07-31 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This study will be an adaptive phase 2/3 investigation. First, 12 subjects will be randomly assigned to receive 1 of the 2 treatment regimens (study drug or placebo) in a 1:1 ratio. After the first 6 subjects have been enrolled and have completed 24 hours post treatment of 2nd dose, the IDMC will review the safety data and will inform whether to continue with staggered enrollment. Randomization ratio for subjects in the following stage will be 1:1. The independent data monitoring committee (IDMC) will review safety data after 12, 24, 48 and 96 patients have been enrolled in each arm. The study will then enroll a total of 121 patients in each arm. An interim analysis will be performed after 80% of recruitment has been reached (n=194). The IDMC will analyze the rate of events in the group under "standard of care".
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A Double-blind, Placebo-controlled, sealed-envelope based. Access to unblinded interim results will be limited to the DMC and unblinded statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Subjects will receive a 1st intravenous dose of 4 mg/kg INM005 (Anti-SARS-CoV-2 hyperimmune equine immunoglobulin F[ab']2 fragments) and a 2nd intravenous dose of 4 mg/kg of INM005. Each dose will be separated by 48 h (± 2 h).
  Interventions: Drug: INM005
- Placebo (Placebo Comparator): Subjects will receive a 1st intravenous dose of Placebo and a 2nd intravenous dose of Placebo. Each dose will be separated by 48 h (± 2 h).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INM005 — The IMP dose to be studied will be 4 mg of protein/kg of subject's weight. The IMP will be added to the 100 mL infusion bag of saline solution. Doses will be administered as an infusion at 2.0 mL/min over 50 min with an interval of 48 h between doses.
  Arms: Active
Drug: Placebo — Placebo substance will be added to the 100 mL infusion bag of saline solution. Doses will be administered as an infusion at 2.0 mL/min over 50 min with an interval of 48 h between doses.
  Arms: Placebo

SUMMARY:
This study aims to analyze the efficacy and safety of passive immunotherapy by administering an equine hyperimmune serum (INM005) against the SARS-CoV2 RBD to Covid19 patients. Improvement of the clinical course 28 days after the start of treatment will be evaluated.

DETAILED DESCRIPTION:
The pandemic caused by the new coronavirus has generated a situation unprecedented in recent history, with several million infected and hundreds of thousands of deaths. This disease is easily transmissible by air. Although a high percentage of cases present mild clinical presentation, approximately 15% of patients present moderate to severe cases and 5% require critical care, with respiratory assistance and a high risk of mortality. No effective therapies for the treatment or prevention of SARS.CoV2 have been identified yet. Preliminary evidence indicates that passive immunotherapy with convalescent plasma could alter the clinical course of this infection in a favorable manner. This strategy, even if confirmed as successful, requires voluntary donation by patients who have recovered, not all of whom are eligible as donors, since the antibody response varies in magnitude in different patients. This adaptive stage II/III study aims to analyze the efficacy and safety of passive immunotherapy by administering a purified Fab fraction of equine hyperimmune serum (INM005) generated from antigenic stimulation with the SARS-CoV2 RBD protein, with the objective of neutralizing the interaction of SARS-CoV-2 with its cellular receptor, thus preventing the multiplication of the virus. The safety of this type of equine hyperimmune sera has already been demonstrated in previous and ongoing protocols with a biologically equivalent product against the E. Coli shiga toxin to treat patients with Hemolytic Uremic Syndrome (CT-INM004-01 and CT-INM004-02). In the present study, eligible patients will with moderate to severe symptoms of COVID-19 that require hospitalization will receive two 4 mg/kg doses of INM005, two days apart, with the aim of improving the clinical course of COVID-19 28 days after the start of treatment with the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of both sexes aged 18 to 79 years of age
2. SARS-CoV-2 infection confirmed by PCR for virus detection
3. Patients with moderate or severe disease by NIH definition, which requires hospitalization.
4. Acceptance to participate in the study by the signature of the informed consent by a subject or their relative, if applicable
5. Be within 10 days of the onset of symptoms at the time of the Screening visit according to a case definition from the National Ministry of Health
6. Female patients of child-bearing age with negative pregnancy test

Exclusion Criteria:

1. Patients who have received treatment with plasma from COVID-19 convalescents.
2. Patients who are participating in other therapeutic clinical trials
3. Patients who require mechanical respiratory assistance or are hospitalized in the ICU at the time of the screening visit.
4. History of anaphylaxis, prior administration of equine serum (por example, anti-tetanus serum or anti-ophidic serum or anti-arachnid toxin serum) or allergic reaction due to contact or exposure to horses.
5. Pregnant or breastfeeding women
6. Patients who, at the doctor's discretion, are likely to die within the next 30 days due to a concomitant disease other than the study disease
7. Patients who are expected to be referred to another institution within 72 hours of enrollment, which prevents proper follow-up of that patient.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Clinical changes in COVID-19 symptoms | 4 weeks
  The primary endpoint will be the proportion of patients who show a change in symptoms 28 days after the administration of the first dose. A responding subject is defined as a subject with improvement in at least 2 categories on the 8-point World Health Organization (WHO) ordinal scale of clinical status or a subject who is discharged.

SECONDARY OUTCOMES:
Pharmacokinetics evaluation of INM005 | 1 week
  INM005 product concentration in serum at different time points after dosing
Time to progression of disease | 4 weeks
  Time to achieve a change in at least 2 categories on the 8-point WHO ordinal scale of clinical status.
  Time to discharge (days). Time to intensive care unit (ICU) discharge (days).
Disease progression | up to 2 weeks
  Proportion of patients who present change in at least 2 categories on the 8-point WHO ordinal scale of clinical status at 7 and 14 days after the start of the treatment.
Discharge | up to 4 weeks
  Proportion of patients discharged at 28 days
Intensive care unit (ICU) hospitalization | up to 4 weeks
  Proportion of patients who require ICU hospitalization
Mechanical ventilation assistance (MVA) | up to 4 weeks
  Proportion of patients who require MVA
Mortality | up to 4 weeks
  Proportion of patients who die due to complications from COVID19
Changes in viral load | up to 3 weeks
  Change in viral load from baseline to 7 and 21 days after the start of the treatment.

OTHER OUTCOMES:
Anti SARS-CoV2 antibodies levels | 3 weeks
  Measurement of anti SARS-CoV2 antibodies titer levels. IgG (0, 21 days)
Changes in Troponin T levels | 3 weeks
  Changes in Troponin T levels will be evaluated at 7 and 21 days as a measurement of disease progression
Changes in D-dimer levels | 3 weeks
  Changes in D-dimer levels will be evaluated at 7 and 21 days as a measurement of disease progression
Changes in Ferritin levels | 3 weeks
  Changes in Ferritin levels will be evaluated at 7 and 21 days as a measurement of disease progression
Changes in LDH levels | 3 weeks
  Changes in LDH levels will be evaluated at 7 and 21 days as a measurement of disease progression
Changes in C-reactive protein levels | 3 weeks
  Changes in C-reactive protein levels will be evaluated at 7 and 21 days as a measurement of disease progression
Immunogenicity | 3 weeks
  Measurement of anti-INM005 antibodies: baseline and 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Sanguineti, Ph.D., Study Director — Inmunova S.A.
Locations (23):
- Argentina (23):
  - Hospital de Cuenca Alta, Cañuelas, Buenos Aires
  - Hospital Prof. Dr. Bernardo A. Houssay, Florida, Buenos Aires
  - Instituto Medico Platense, La Plata, Buenos Aires
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Hospital Municipal Emilio Zerboni, San Antonio de Areco, Buenos Aires
  - Hospital Alta Complejidad "El Cruce" Dr. Néstor Carlos Kirchner, San Juan Bautista, Buenos Aires
  - Hospital Municipal Dr. Diego E. Thompson, San Martín, Buenos Aires
  - Hospital Pablo Soria, San Salvador de Jujuy, Jujuy Province
  - Hospital Provincial Neuquén "Dr. Eduardo Castro Rendón", Neuquén, Neuquén Province
  - Hospital Centro de Salud Zenón J. Santillán, San Miguel de Tucumán, Tucumán Province
  - Sanatorio Guemes, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Muñiz, Buenos Aires
  - Hospital Pirovano, Buenos Aires
  - Centro Gallego de Buenos Aires, Ciudad Autonoma de Buenos Aire
  - Clínica Adventista Belgrano, Ciudad Autonoma de Buenos Aire
  - Clínica Pasteleros, Ciudad Autonoma de Buenos Aire
  - Clínica Zabala, Ciudad Autonoma de Buenos Aire
  - Fundación Favaloro, Ciudad Autonoma de Buenos Aire
  - Hospital Español de Buenos Aires, Ciudad Autonoma de Buenos Aire
  - Hospital G. A. Carlos G. Durand, Ciudad Autonoma de Buenos Aire
  - Sanatorio Agote, Ciudad Autonoma de Buenos Aire
  - Sanatorio Sagrado Corazón, Ciudad Autonoma de Buenos Aire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] Lopardo G, Belloso WH, Nannini E, Colonna M, Sanguineti S, Zylberman V, Munoz L, Dobarro M, Lebersztein G, Farina J, Vidiella G, Bertetti A, Crudo F, Alzogaray MF, Barcelona L, Teijeiro R, Lambert S, Scublinsky D, Iacono M, Stanek V, Solari R, Cruz P, Casas MM, Abusamra L, Luciardi HL, Cremona A, Caruso D, de Miguel B, Lloret SP, Millan S, Kilstein Y, Pereiro A, Sued O, Cahn P, Spatz L, Goldbaum F; INM005 Study Group. RBD-specific polyclonal F(ab )2 fragments of equine antibodies in patients with moderate to severe COVID-19 disease: A randomized, multicenter, double-blind, placebo-controlled, adaptive phase 2/3 clinical trial. EClinicalMedicine. 2021 Apr;34:100843. doi: 10.1016/j.eclinm.2021.100843. Epub 2021 Apr 11. PMID 33870149